CLINICAL TRIAL: NCT00741481
Title: Evaluation of Prognostic and Predictive Value of PETSCAn in ColoRectal Cancer (CRC)
Brief Title: PET Evaluation of Response After 1 Course of Chemotherapy as Predictor of Treatment Outcome.
Acronym: earlyPETmCRC
Status: Completed | Type: Observational
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Alain Hendlisz, MD, Head, Gastroenterology Unit, Institut Jules Bordet, Service de Medecine
Other Study IDs: earlyPETmCRC; comité éthique IJB n° 1377
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Colorectal Cancer Metastatic; Early Response Evaluation; Fdg-PET
Keywords: metastatic colorectal cancer; fdg pet; response evaluation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: all study population
  Interventions: Procedure: FDG-PET imaging

INTERVENTIONS:
Procedure: FDG-PET imaging — FDG-PET imaging at D0 and D14 of first course of a new chemotherapy for advanced colorectal cancer
  Other Names: PET-CT SCan

SUMMARY:
Study hypothesis : early decrease in fdg-pet measured SUV max after 1 cycle of chemotherapy can accurately predict response of chemotherapy as assessed by conventional radiology after 3 cycles of chemotherapy.

FDG-PET imaging will be done at J0 and J14 of a new line of chemotherapy treatment in metastatic colorectal cancer.

SUV max will be recorded and delta SUVmax will be compared to the results of conventional radiological evaluation after 3 courses of chemotherapy. Results will also be compared to the time to disease progression.

DETAILED DESCRIPTION:
statistical hypothesis : Sample size calculation for FDG-PET in metastatic patients.

In the paper of Cascini et al. [1], they have 18 patients with a TRG response (TRG = Tumor Regression Grade) and 15 patients with no response.

SUV mean was measured at baseline and at day 12 in all 33 patients. All 33 patients showed a reduction in SUV-mean from baseline to day 12. The median reduction in SUV-mean was 63% (mean 66%) in responding tumors and 22% (mean 22%) for non responding tumors. Using a cutoff level of 52% a perfect accuracy could be obtained, i.e. all responding tumors had a SUV-mean reduction higher than 52% and all non responding tumors had a SUV-mean reduction lower than 52%.

(Standard deviation of the SUV-mean reduction was 25.) All 33 patients showed also a reduction in SUV-max from baseline to day 12. The median reduction in SUV-max was 62% in responding tumors and 28% in non responding tumors. (No information about mean or standard deviation of SUV-max available in [1].) Based on the data of SUV-mean we can do a power calculation based on the Wilcoxon test: In order to demonstrate an absolute difference in the mean of ΔSUV-mean of 44% between responding and non responding patients, with an estimated standard deviation of 25, using 35 patients (50% response, 50% no response), at a significance level of 5%, we obtain a power of 0.98.

For SUV-max, if we assume that the difference in the means is similar to the difference in the medians, i.e. 34% and the standard deviation is similar to the one of SUV-mean, i.e. 25, we obtain a power of 0.93 If we, to be safe, are a little bit less optimistic and estimate that the difference in the mean of ΔSUV-max between responding and non responding tumors would be a little lower than in [1]: 35%, and the standard deviation a little bit higher: 30, then we need 40 patients at a power of 0.90

Référence 1 : Cascini GL, Avallone A, Delrio P, Guida C, Tatangelo F, Marone P et al.: F-18-FDG PET is an early predictor of pathologic tumor response to preoperative radiochemotherapy in locally advanced rectal cancer. Journal of Nuclear Medicine 2006, 47: 1241-1248.

ELIGIBILITY:
Inclusion Criteria:

* advanced colorectal cancer
* evaluable disease
* signed informed consent

Exclusion Criteria:

* no other cancer
* no other life-threatening condition
* unwillingness or inability to sign informed consent
* active cerebral metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 yrs old advanced evaluable colorectal cancer beginning a new line of chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2006-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
compare fdg-pet variations after 1 course of chemotherapy to chemotherapy outcome measured by time to disease progression | Time to Disease progression

SECONDARY OUTCOMES:
compare fdg-pet variations after 1 course of chemotherapy to chemotherapy outcome measured by tumour response rate following RECIST criteria. | response rate

CONTACTS AND LOCATIONS:
Overall Officials: Alain - Hendlisz, MD, Principal Investigator — Institut Jules Bordet, Université Libre de Bruxelles, Brussels
Locations (1):
- Institut Jules Bordet, Université Libre de Bruxelles, Brussels, Belgium